CLINICAL TRIAL: NCT00680654
Title: Interaction Study to Investigate Safety, Tolerability, Pharmacokinetics and the Impact on Pulmonary and Systemic Hemodynamics of Single Doses of 0.5 and 1 mg of BAY 63-2521 in Patients With PAH and Stable Treatment of Sildenafil 20 mg TID in a Non-randomized, Non-blinded Design
Brief Title: Interaction Study in Patients With Pulmonary Hypertension and Stable Treatment of Sildenafil 20 mg TID
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11917; 2008-000914-65 (EudraCT Number)
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — The investigational drug will be given twice per subject, as single dose administration of BAY 63-2521 (0.5 mg and 1.0 mg) during the hemodynamic investigation.

SUMMARY:
This study is to demonstrate the safety, tolerability, pharmakokinetic and pharmacodynamic effect of BAY63-2521 in patients with pulmonary hypertension and stable treatment of sildenafil 20 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary hypertension stable for the last 6 weeks
* Treated with Sildenafil 3 × 20 mg
* Undergoing routine invasive diagnostics.

Exclusion Criteria:

* Pre-existing lung disease other than pulmonary arterial hypertension,
* Acute or severe chronic left heart failure,
* Severe coronary artery disease,
* Uncontrolled arterial hypertension;
* Congenital or acquired valvular or myocardial disease except acquired tricuspid valve insufficiency due to pulmonary hypertension,
* Systolic blood pressure < 100 mmHg, heart rate < 55 bpm or >105 bpm, PaO2/FiO2 < 50 mmHg,
* PaCO2 > 55 mmHg,
* Severe hepatic insufficiency,
* Severe renal insufficiency,
* Administration of strong CYP3A4 inhibitors or inductors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Impact of a single dose of BAY63-2521 on pharmacodynamic parameters of the pulmonary system, on safety, tolerability and pharmacokinetics. | At baseline, throughout study days 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Germany (5):
  - Heidelberg, Baden-Wurttemberg
  - Löwenstein, Baden-Wurttemberg
  - Giessen, Hesse
  - Greifswald, Mecklenburg-Vorpommern
  - Dresden, Saxony

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/